CLINICAL TRIAL: NCT06101472
Title: Rotational Stability and Clinical Response of the ASQELIO Toric Biaspheric Monofocal Lens.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: AST Products, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ASQM022023
Record Dates: First submitted 2023-09-20; First posted 2023-10-26 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2023-10

CONDITIONS: Cataract
Keywords: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pseudophakic subjects implanted with the ASQELIO toric IOL: Adult subjects undergoing cataract surgery by routine clinical practice with ASQELIO Toric Biaspheric Monofocal Lens in at least one eye.
  Interventions: Device: ASQELIO Toric Biaspheric Monofocal Lens

INTERVENTIONS:
Device: ASQELIO Toric Biaspheric Monofocal Lens — Intraocular lens implantation in cataract surgery

SUMMARY:
The goal of this observational study is to evaluate the rotational stability and clinical performance of the ASQELIO Toric lens in candidates for cataract surgery with ASQUELIO Toric intraocular lens (IOL) implantation.

Information will be obtained from patients operated by routine clinical practice with toric monofocal ASQELIO IOL in at least one eye. After confirmation of inclusion, the preoperative examination will be performed, and after surgery an evaluation will be performed the following day, one week, one month and three months after surgery.

DETAILED DESCRIPTION:
In cataract surgery, the opacified lens is removed by phacoemulsification and replaced by an artificial IOL.The most common risk of cataract surgery is the development of a condition called posterior capsular opacification (PCO) that causes further deterioration of visual function. Toric intraocular lenses correct corneal astigmatism and avoid residual refractive errors in these subjects. For their efficacy in this refractive error correction, it is essential that, once implanted, these lenses are rotationally stable.The goal of this observational study is to evaluate the rotational stability and clinical performance of the ASQELIO Toric lens during the first 3 months after implantation.

All patients participating in the study are candidates for cataract surgery with ASQUELIO Toric intraocular lens (IOL) implantation model TLIO130 from AST Products, Inc., with CE marking.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 22 years of age or older undergoing cataract surgery in at least 1 eye and implanted with LIO ASQELIO.
* Subjects for whom postoperative emmetropia was planned (±0.5 D spherical equivalent)

Exclusion Criteria:

* Preoperative corneal astigmatism less than 0.75D
* Patients who do not provide informed consent
* Patients who do not understand the study procedure.
* Previous corneal surgery or trauma.
* Irregular cornea (e.g. keratoconus).
* Microphthalmos.
* Severe corneal dystrophy.
* Pregnant or breastfeeding'.
* Rubella
* Mature/dense cataract making eye bottom preoperative examination difficult.
* Previous retinal detachment.
* Concurrent participation in other research with drugs or clinical devices.
* Expect to require another eye surgery during the study period.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects who are candidates for cataract surgery and implantation of toric monofocal ASQELIO IOL in at least one of their eyes.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Rotational stability of the implant | During 3 months after IOL implantation
  Evaluated at each visit by analysis of slit-lamp backlight images, following the method described by Wolffsohn and Buckhurst. By means of backlighting, the IOL markings indicating the axis in which the astigmatic power is located will be observed and by image analysis it will be determined and quantified whether the lens has been rotated.
Visual acuity | During 3 months after IOL implantation
  Best corrected distance visual acuity in LogMAR units using the ETDRS chart

SECONDARY OUTCOMES:
Refraction | During 3 months after IOL implantation
  Using subjective refraction methods.
Adverse events | During 3 months after IOL implantation
  Adverse events are obtained from solicited and spontaneous comments from the subjects and from observations made by the investigator.
Satisfaction and quality of vision questionnaire | During 3 months after IOL implantation
  Collected from solicited and spontaneous comments from the subjects, as well as the Catquest-9SF questionnaire, validated in Spanish.
  The subjective assessment of the quality of vision will be determined by an additional questionnaire about the presence of visual symptoms related to positive dysphotopsias (halos, glare and glare).

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Tañá, Dr, Principal Investigator — Oftalmología Vistahermosa SL
Locations (3):
- Spain (3):
  - Oftalvist Alicante, Alicante
  - OftalVist Madrid, Madrid
  - OftalVist Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No